CLINICAL TRIAL: NCT06885463
Title: The Role of Platelets Rich Plasma Combined With PDO Threads in Treatment of Stress Incontinence in Egyptian Women
Brief Title: PRP & PDO Threads in Treatment of Stress Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asem Anwar Moussa, Professor, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00000501
Record Dates: First submitted 2025-03-12; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Stress Incontinence, Female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- platelets rich plasma combined with PDO threads (Experimental)
  Interventions: Procedure: platelets rich plasma combined with PDO threads

INTERVENTIONS:
Procedure: platelets rich plasma combined with PDO threads — 1. Injections of platelets-rich plasma in the Anterior Vaginal Wall.
  2. PDO thread placement in the paraurethral, lateral urethrovaginal, and suburethral areas

SUMMARY:
The study will include 10 women with pure or predominant SUI symptoms, with severe urodynamic stress incontinence on urodynamics defined as loss of urine with sudden increases in abdominal pressure: eg, coughing, sneezing, or laughing). This will be conducted at the Department of Obstetrics and Gynecology, Faculty of Medicine, Al-Azhar University. The purpose of study is to evaluate the efficacy and safety of platelets rich plasma combined with PDO threads in the treatment of stress incontinence in Egyptian women.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant Women with SUI
* Age between 20 to 45 years
* Patients had a history of failed conservative treatment
* Patients were on the waiting list for surgical treatment of SUI

Exclusion Criteria:

* Under anti-platelet agent treatment
* Under NSAIDs
* Platelet dysfunction syndrome
* Critical thrombocytopenia
* Hypofibrionogenaemia
* Sepsis
* Acute and chronic infections
* Chronic liver disease
* Anti-coagulation therapy
* History of malignancy
* Pregnancy
* history of active malignant pathology
* mental disorders making them unable to give consent
* genitourinary fistula
* pelvic organs prolapse stage >2 according to the Pelvic Organ Prolapse Quantification system, and detrusor overactivity on urodynamics.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
evaluation of reported SUI symptoms | After 4 months
  subjective evaluation of reported SUI symptoms, indicated by the patient's response to question of the ICIQ-FLUTS questionnaire: "Does urine leak when you are physically active, exert yourself, cough or sneeze?"

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Al-Azhar University., Cairo, Egypt